CLINICAL TRIAL: NCT04244942
Title: CERAMENT™| Bone Void Filler Device Registry
Status: Recruiting | Type: Observational
Sponsor: BONESUPPORT AB (Industry)
Responsible Party: Sponsor
Other Study IDs: S025/2018
Record Dates: First submitted 2020-01-15; First posted 2020-01-28 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: CERAMENT BVF — CERAMENT BONE VOID FILLER is a synthetic biphasic bone graft substitute.

SUMMARY:
A device registry to compile data on the performance of CERAMENT BONE VOID FILLER in normal use.

DETAILED DESCRIPTION:
A device registry to compile data on the performance of CERAMENT BONE VOID FILLER in normal use.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over (on the day of surgery)
* Receive CERAMENT BVF as a component of their treatment at a participating, contracted center or healthcare provider, in accordance with the IFU for the implanted product
* In receipt of patient information leaflet and have signed appropriately designed informed consent

Exclusion Criteria:

* Any exclusion criteria as per IFU for CERAMENT BVF
* Any off-label use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The racial, gender, and ethnic characteristics of the individuals approached for participation in this Observational Registry Study shall reflect the demographics of patients that would ordinarily received CERAMENT BVF for the treatment of their condition at the designated investigative centers. No individuals shall be excluded from participation in the Observational Registry Study based on race, nationality, ethnicity, gender or sexuality.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-03-30 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Unexpected device performance will be collected as they occur at time of surgery and on an ongoing basis thereafter, with formal scheduled review at 12 and 18 months | 12 months
  Unexpected device performance will be collected as they occur at time of surgery and on an ongoing basis thereafter, with formal scheduled review at 12 and 18 months
Unexpected device performance will be collected as they occur at time of surgery and on an ongoing basis thereafter, with formal scheduled review at 12 and 18 months | 18 months
  Unexpected device performance will be collected as they occur at time of surgery and on an ongoing basis thereafter, with formal scheduled review at 12 and 18 months
Complaints will be collected as they occur at time of surgery and on an ongoing basis thereafter, with formal scheduled review at 12 and 18 months | 12 months
  Complaints will be collected as they occur at time of surgery and on an ongoing basis thereafter, with formal scheduled review at 12 and 18 months
Complaints will be collected as they occur at time of surgery and on an ongoing basis thereafter, with formal scheduled review at 12 and 18 months | 18 months
  Complaints will be collected as they occur at time of surgery and on an ongoing basis thereafter, with formal scheduled review at 12 and 18 months
Adverse events will be collected as they occur at time of surgery and on an ongoing basis thereafter, with formal scheduled review at 12 and 18 months | 12 and 18 months
  Adverse events will be collected as they occur at time of surgery and on an ongoing basis thereafter, with formal scheduled review at 12 and 18 months
Adverse events will be collected as they occur at time of surgery and on an ongoing basis thereafter, with formal scheduled review at 12 and 18 months | 12 months
  Adverse events will be collected as they occur at time of surgery and on an ongoing basis thereafter, with formal scheduled review at 12 and 18 months
adverse device events will be collected as they occur at time of surgery and on an ongoing basis thereafter, with formal scheduled review at 12 and 18 months | 18 months
  Adverse device events will be collected as they occur at time of surgery and on an ongoing basis thereafter, with formal scheduled review at 12 and 18 months
SAEs will be collected as they occur at time of surgery and on an ongoing basis thereafter, with formal scheduled review at 12 and 18 months | 12 months
  SAEs will be collected as they occur at time of surgery and on an ongoing basis thereafter, with formal scheduled review at 12 and 18 months
SAEs will be collected as they occur at time of surgery and on an ongoing basis thereafter, with formal scheduled review at 12 and 18 months | 18 months
  SAEs will be collected as they occur at time of surgery and on an ongoing basis thereafter, with formal scheduled review at 12 and 18 months

SECONDARY OUTCOMES:
Radiological assessment at 6 and 12 months. Objective assessment of regeneration | 6 Months
  Bone healing
Radiological assessment at 6 and 12 months. Objective assessment of regeneration | 12 Months
  Bone healing
Pain VAS score | 6, 12, and 18 Months
  Pain assessment at 6,12, and 18 months
EQ-5D-3L | 6, 12, and 18 months
  Functional assessment at 6, 12, and 18 months

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - HonorHealth, Scottsdale, Arizona
  - Golden Orthopedic Knee, Hip, Shoulder and Foot Center, Boca Raton, Florida
  - Sports and Orthopedic Center, Boca Raton, Florida
  - Dr. Peter Merkle, Pompano Beach, Florida
  - Florida Orthopedic Foot & Ankle Center, Sarasota, Florida
  - James Cottom, Sarasota, Florida
  - Indiana University, Indianapolis, Indiana
  - OrthoIndy, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Research Foundation of The State University of New York, Syracuse, New York
  - OrthoCarolina, Charlotte, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No